CLINICAL TRIAL: NCT06585475
Title: The Effectiveness of Structured Training According to the Premenstrual Syndrome Symptom Map
Brief Title: Investigation of the Effectiveness of Structured Education According to Premenstrual Syndrome Symptom Map
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 23.08.2024
Record Dates: First submitted 2024-09-03; First posted 2024-09-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Premenstrual Syndromes; Education; Menstrual Cycle Disorder
Keywords: life satisfaction; pain; depression; stress; anxiety
MeSH Terms: conditions — Premenstrual Syndrome; Menstruation Disturbances; Personal Satisfaction; Pain; Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The intervention group received a 3-session PMS symptom map-structured training by the responsible and first author (ADK). Before the training, pre-test data were collected using data collection tools (VAS pain scoring, DAS depression stress anxiety assessment scale, premenstrual syndrome assessment scale and premenstrual syndrome-specific life satisfaction scale). After the training, post-test data were collected on the last day of the 1nd cycle.
  Interventions: Behavioral: Structured training according to premenstrual syndrome symptom map
- Control group (No Intervention): No intervention was applied to the control group. After the participants were divided into groups by randomization, pre-test data were collected using data collection tools (VAS pain scoring, DAS depression stress anxiety rating scale, premenstrual syndrome rating scale and premenstrual syndrome specific life satisfaction scale). After the pre-test, post-test data were collected on the last day of the cycle after 1 menstrual cycles.

INTERVENTIONS:
Behavioral: Structured training according to premenstrual syndrome symptom map — A symptom map consisting of evidence-based practices for coping with PMS symptoms was created. An educational content based on this map was prepared and applied to women with PMS to evaluate whether it was effective compared to the control group.
  Arms: Experimental group

SUMMARY:
In this study, it was aimed to evaluate the effectiveness of the training structured according to the PMS symptom map. This experimental (randomised-controlled) study was conducted with women of reproductive age with PMS. Women who met the inclusion criteria and volunteered to participate in the study constituted the sample of the study. As a result of block randomisation, 55 women were assigned to the intervention group and 55 women to the control group. Pre-test data were collected from the women allocated to the intervention and control groups by means of data collection tools (VAS pain scoring, DAS depression stress anxiety assessment scale, Premenstrual syndrome assessment scale and premenstrual syndrome-specific life satisfaction scale). The intervention group received a 3-session structured training according to the PMS symptom map, while the control group did not receive any intervention. Women in the intervention group completed the post-test data on the last day of the 2nd cycle after the training, while women in the control group completed the post-test data on the last day of the 2nd cycle after the pre-test.

ELIGIBILITY:
Inclusion Criteria:

Meeting ACOG's PMS diagnostic criteria Being over 18 years of age, Not using psychotherapeutic medications, Not having a mental illness, Not being pregnant, Agreeing to participate in the study

Exclusion Criteria:

Not having regular menstruation in the last 3 months, Using analgesics during menstruation while participating in the study.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 101 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-08-05 (Actual)

PRIMARY OUTCOMES:
Premenstrual syndrome assessment scale | pre-intervention, 2 month after intervention
  a scale used to measure the degree of premenstrual syndrome
premenstrual syndrome specific life satisfaction scale | pre-intervention, 2 month after intervention
  Premenstrual syndrome specific life satisfaction scale evaluates life satisfaction of women with PMS
DAS depression stress anxiety assessment scale | pre-intervention, 2 month after intervention
  DAS depression stress anxiety assessment scale, evaluates psychological symptoms
VAS pain score | pre-intervention, 2 month after intervention
  1.421 / 5.000 VAS pain score measures pain score

CONTACTS AND LOCATIONS:
Locations (1):
- Sakarya University, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No